CLINICAL TRIAL: NCT05163899
Title: Phase II Pilot Randomized-Controlled Trial for the Investigation of the Preliminary Efficacy of Surgical Sectioning of the Filum Terminale in Treating Occult Tethered Cord Syndrome Patients
Brief Title: Investigation of Surgical Sectioning of the Filum Terminale in Treating Occult Tethered Cord Syndrome Patients
Acronym: OCCULT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-06022262
Record Dates: First submitted 2021-11-08; First posted 2021-12-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Tethered Cord; Tethered Cord Syndrome; Occult Spina Bifida; Spina Bifida Occulta
Keywords: tethered cord; occult; filum terminale; tight filum
MeSH Terms: conditions — Spinal Cord Injuries; Neural Tube Defects; Spina Bifida Occulta | interventions — Laminectomy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two arms: surgical untethering or medical management only. Symptom improvement and adverse events will be assessed and recorded for 1 year from initiation of treatment. After a minimum of 1 year, subjects who were randomized to the medical management arm may cross over to the surgical arm if the PI deems it is in the subject's best interest to do so.
Who Masked: Outcomes Assessor
Masking Description: For a surgical vs non-surgical trial, the investigator can not be masked thus only the evaluators will be unaware of the arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Filum release
  Interventions: Procedure: Release of filum terminale
- Observation (No Intervention): Medical Management only

INTERVENTIONS:
Procedure: Release of filum terminale — Surgery will be offered to section the filum terminale
  Other Names: Laminectomy for tethered cord release
  Arms: Surgery

SUMMARY:
The investigators hypothesize that surgical release of the filum terminale (strand of fibrous tissue at the end of the spinal cord) is a more efficacious treatment option for symptomatic relief than medical management in subjects with Occult Tethered Cord Syndrome (OTCS) and that the risks do not outweigh the benefit profile.

DETAILED DESCRIPTION:
This is a phase II pilot randomized-controlled, single-site trial to determine if surgical untethering of the filum terminale is more effective, preliminarily, than medical management as a treatment option for OTCS. Subjects will be randomized to one of two arms: surgical untethering or medical management only. Symptom improvement and adverse events will be assessed and recorded for 1 year from initiation of treatment. After a minimum of 1 year, subjects who were randomized to the medical management arm may cross over to the surgical arm if the PI deems it is in the subject's best interest to do so. The exploratory hypothesis is that surgery for OTCS is both safe and more effective than medical management at relieving the symptoms of OTCS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 2 and < 80 years of age.
* Refractory to medical management of symptoms for at least 1 year.
* Documentation of OTCS, as defined by a total score of at least 30 on the following scale:

OCCULT Grading Scale (Score 0-100) Orthopedic Abnormality: 0-15; Central Nervous System Dysfunction: 0-25; Cutaneous Stigmata: 0-10; Urological or Bowel Dysfunction: 0-25; Lumbosacral Anatomy: 0-15; Tissue Integrity Disorder: 0-10.

Exclusion Criteria:

* Subjects < 2 or > 80 years of age.
* Radiographically identified tethered cord, as defined by any of the following:

  * A low-lying conus (at or below the L2-3 disc space)
  * A thickened filum (>2 mm)
  * Fat in the filum or lipoma
  * Distinct adhesion or tethering.
* A history of Meningocele manqué or Myelomeningocele.
* Cutaneous markings of dermal sinus tract.
* History of prior surgery on the lumbar spine.
* History of prior surgery for spinal dysraphism.
* History of prior infection or autoimmune condition of the central nervous system.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms related to tethered cord, as measured by the OCCULT Scale | Baseline, 1 year
  Combination of neurologic, urologic, orthopedic, and cutaneous assessments. The OCCULT Scale is from 0-100, with 0 being none of the listed signs/symptoms present and 100 being all listed signs/symptoms present with maximum severity.

SECONDARY OUTCOMES:
Change in urologic incontinence score | Baseline, 1 year
  Score is measured by the International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form. The minimum score is 0 and the maximum score is 21. The higher the score, the more severe the urinary incontinence symptoms and/or effect of symptoms on quality of life.
Change in fecal incontinence score | Baseline, 1 year
  Score is measured by the Rapid Assessment Faecal Incontinence Score. The minimum score is 0 and the maximum score is 20. The higher the score, the more severe the fecal incontinence symptoms and/or effect of symptoms on quality of life.
Number of patients who cross over | 1 year
Percent of patients with a decrease in anticholinergic medications at 1 year post-surgery | 1 year
  For patients who presented with urological symptoms
Number of intra-operative findings that are discordant with MRI interpretations | Intraoperative
  To examine whether there is a limitation in MRI in identifying pathology that is identified at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Greenfield, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michael MM, Garton ALA, Kuzan-Fischer CM, Uribe-Cardenas R, Greenfield JP. A critical analysis of surgery for occult tethered cord syndrome. Childs Nerv Syst. 2021 Oct;37(10):3003-3011. doi: 10.1007/s00381-021-05287-5. Epub 2021 Jul 15. PMID 34268593